CLINICAL TRIAL: NCT06223256
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of NBL-028 in Patients With Advanced Solid Tumors
Brief Title: A Study of NBL-028 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NovaRock Biotherapeutics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBL-028-001
Record Dates: First submitted 2023-12-18; First posted 2024-01-25 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NBL-028 (Experimental): Patients will be treated with NBL-028 at starting dose of 0.01 mg/kg in dose escalation stage. In dose expansion stage, patients will be treated with NBL-028 at the recommended dose or multiple doses (if necessary) determined in the dose escalation stage.
  Interventions: Drug: NBL-028

INTERVENTIONS:
Drug: NBL-028 — Intravenous infusion (IV), once every two weeks (one treatment cycle is 4 weeks).

SUMMARY:
This is a multi-center, single agent study conducted in patients with advanced solid tumor types known to express Claudin 6 (CLDN6) for whom standard of care therapies are not available, are no longer effective, or not tolerated. This study consists two stages: dose-escalating and dose-expansion.

Dose escalation will be guided by the Bayesian optimal interval (BOIN) design including accelerated titration to determine the maximum tolerated dose (MTD) of NBL-028. Dose expansion - Additional patients (no more than 200) will be enrolled at the recommended dose or multiple doses (if necessary) determined in the dose escalation stage. Sponsor may elect to enroll specific tumor types into four cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old, should have fully understood the study and voluntarily signed an informed consent form.
2. Patients with pathologically diagnosed advanced solid tumors with positive expression of CLDN6. Stage I: Patients have failed or cannot tolerate standard of care, or without standard treatment; Stage Ⅱ: Previously treated advanced solid tumors.
3. Be able to provide previously well-preserved tumor tissue sections, or agree to undergo tumor tissue biopsy for central laboratory biomarker testing.
4. At least one measurable target lesion according to RECIST 1.1.
5. ECOG performance status of 0 or 1 at screening.
6. Life expectancy ≥3 months.
7. Adequate organ function within 7 days prior to the first dose defined as: Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥100×10^9/L;. Hemoglobin (HGB) ≥90 g/L; Serum creatinine ≤ 1.5 × ULN or Calculated creatinine clearance (CrCl) (Cockcroft-Gault formula) ≥50 mL/min; Total bilirubin (TBIL) ≤1.5×ULN (≤3×ULN when patients with Gilbert's disease); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN if liver involvement is known).
8. Serum pregnancy test for women of childbearing potential (WOCBP) is negative within 7 days prior to the first dose of the investigational drug. The patient and his/her spouse must agree to use adequate contraception from signing of informed consent form (ICF) to 3 months after the last dose, during which women should be non-lactating and men should refrain from donating sperm.

Exclusion Criteria:

1. Previously received CLDN6-targeted or CD137-targeted treatment.
2. Known uncontrolled central nervous system (CNS) cancer including CNS metastasis, meningeal metastasis, or spinal cord compression.
3. Patients with high risk of bleeding due to tumor invasion of important arteries.
4. Has uncontrolled serous cavity effusion (such as pleural effusion, abdominal effusion, or pericardial effusion, etc) requiring repeated drainage.
5. Has adverse events due to previous anti-tumor treatments that have not yet recovered to ≤Grade 1 according to NCI-CTCAE v5.0;
6. Developed immune-related adverse events (irAE) of grade ≥3 (CTCAE 5.0) with prior immunotherapy
7. Known to exist any other malignant tumor requiring intervention.
8. Have received anti-tumor treatments (such as chemotherapy, targeted therapy, biological therapy, etc.) or any other investigational drugs or treatments within 4 weeks or 5 half-lives, whichever is shorter.
9. Have received a live viral vaccine within 4 weeks before the first dose of study drug.
10. Have received immunosuppressive medications within 2 weeks prior to the first dose of study drug.
11. Have active or serious bacterial, fungal, or viral infection requiring systemic anti-infective treatment within 2 weeks prior to the first dose of study drug.
12. Have received radiation therapy or other localized palliative treatment within 2 weeks before the first dose of study drug.
13. Have undergone major surgery within 4 weeks before the first dose of study drug, or scheduled to have major surgery during the study.
14. Have a history of serious cardiovascular disease.
15. Have active or history of autoimmune diseases.
16. A history of immunodeficiency, including HIV testing positive, or having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.
17. Active hepatitis B; hepatitis C infection; syphilis infection, active tuberculosis.
18. Hypersensitive to humanized monoclonal antibody products.
19. Women during lactation or pregnancy.
20. Any male and female patients with fertility who refuse to use effective contraceptive methods throughout the entire trial period and within six months after the last administration.
21. Other conditions that, in the opinion of the investigator, may affect the safety or compliance of drug treatment in this study, including but not limited to: psychiatric disorders, any severe or uncontrollable diseases, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | Up to approximately 1 years
  Dose-limiting toxicity
Incidence and severity of adverse events (AE) and serious adverse events (SAE) Incidence, nature, and severity of adverse events will be graded according to the NCI CTCAE v5.0 | Up to approximately 3 years
  adverse events (AEs) and severe adverse events (SAEs)
Maximum Tolerated Dose（MTD） of NBL-028 | Up to approximately 1 years
  Maximum Tolerated Dose
Recommended Phase 2 dose（RP2D） | Up to approximately 1 years
  Recommended Phase 2 dose

SECONDARY OUTCOMES:
Overall response rate (ORR).Determined using RECIST v1.1 criteria. | Up to approximately 3 years
  Objective response rate
Pharmacokinetic (PK) profile of YBL-006.Assessed by parameter Cmax. | Up to approximately 3 years
  Observed maximum concentration
Pharmacokinetic (PK) profile of YBL-006.Assessed by parameter Area under curve（AUC）. | Up to approximately 3 years
  AUC0-t
Pharmacokinetic (PK) profile of YBL-006.Assessed by parameter Tmax. | Up to approximately 3 years
  Time to maximum concentration
Pharmacokinetic (PK) profile of YBL-006.Assessed by parameter t1/2. | Up to approximately 3 years
  Apparent terminal Half-Life
anti-drug antibody（ADA） | Up to approximately 3 years
  anti-drug antibody titer
Disease control rate（DCR） | Up to approximately 3 years
  Disease control rate
Duration of response (DoR) | Up to approximately 3 years
  Duration of response
Progression free survival（PFS） | Up to approximately 3 years
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Ph.D, Principal Investigator — Sun Yat-Sen University (SYSU) Cancer Center
Locations (1):
- No.896 East Zhongshan Road, Shijiazhuang, Hebei Province, China., Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No